CLINICAL TRIAL: NCT00606229
Title: A Multicenter Investigative Study of the Safety and Efficacy of Long-term Administration of Aripiprazole in Combination With Mood Stabilizer for the Treatment of Patients With Bipolar Disorder Experiencing a Manic or Mixed Episode
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031-07-001
Record Dates: First submitted 2008-01-19; First posted 2008-02-01 (Estimated); Results first posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — oral, 24mg/day
  Other Names: OPC-14597

SUMMARY:
To assess the safety and efficacy of long-term administration of aripiprazole in combination with mood stabilizer (lithium or valproate) in an unblinded manner in patients with Bipolar I Disorder experiencing a manic or mixed episode

ELIGIBILITY:
Inclusion Criteria:

* Trial subjects will be men and women of age 18 or above and below the age of 65 who will not be turning 65 during the trial.
* Patients have the ability to understand and to provide informed consent to the examination, observation, and evaluation processes specified in this protocol, and have signed the informed consent form based on a full understanding of the trial.
* Patients who meet DSM-IV-TR criteria for manic or mixed episodes and have been diagnosed as having "296.4x Bipolar I Disorder in which the most recent episode was manic" or "296.6x Bipolar I Disorder in which the most recent episode was mixed"
* Patients with a YMRS total score of 16 or more

Exclusion Criteria:

* Patients presenting with a clinical picture and/or history that is consistent with a DSM-IV-TR diagnosis of:

  * Delirium, dementia, amnestic disorder, or other cognitive disorders
  * Schizophrenia or other psychotic disorder
  * Personality disorder
* Patients experiencing their first manic or mixed episode
* Patients whose current manic episode has lasted for more than 4 weeks
* Patients with psychotic symptoms that are clearly due to another general medical condition or direct physiological effects of a substance
* Patients who have met DSM-IV-TR criteria for a substance-related disorder within 3 months (90 days) prior to informed consent (excluding caffeine- and nicotine-related disorders, but including abuse of benzodiazepines)
* Patients who have received ECT treatment within 8 weeks prior to informed consent
* Patients who are expected to require administration of ultrashort-acting or short-acting benzodiazepine receptor agonist hypnotics and antianxiety drugs (See (1) of 4.2.2) at doses exceeding the equivalent of 15 mg/day of diazepam (Only for those patients using such drugs)
* Patients at significant risk of developing a severe adverse event. Patients who have a medical condition that would interfere with assessments of safety or efficacy during the course of the trial, or who have a history of such a condition.
* Patients who have received any of the following treatments during the screening period

  * Reserpine
  * Levodopa, dopamine receptor stimulants
  * Monoamine oxidase inhibitors
  * Psychostimulants
  * Thyroid hormones, antithyroid drugs
  * Corticosteroids (other than topical preparations)
  * Adrenaline
  * All other investigational or unapproved agents
  * ECT
  * Light therapy
* Patients judged to have a diabetic blood glucose level (judgment based on use of a self-monitoring blood glucose meter permissible), or patients whose HbA1c is 6.5% or higher
* Patients with a history or a complication of diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Department of Clinical Research and Development, Division of New Product Evaluation and Development
Locations (5):
- Japan (5):
  - Chugoku Region
  - Hokuriku Region
  - Kanto Region
  - Kinki Region
  - Shikoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: Twenty-four milligrams of aripiprazole (four 6-mg tablets) were administered orally once daily for 24 weeks (168 days) in an unblinded manner. The dose could be increased to a maximum of 30 mg/day (five 6-mg tablets).
Period: Overall Study
Arm/Group | Aripiprazole
Started | 41
Completed | 19
Not Completed | 22
Not completed — Adverse Event | 11
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 4
Not completed — does not meet inclusion criterion 1-3 | 4
Not completed — change of residence or other commitments | 2

BASELINE CHARACTERISTICS:
Population: Results obtained from the LOCF dataset of 40 subjects of the Full Analysis Set (FAS) (excluding 1 subject whose post-dose data of efficacy endpoint were not available from the 41 treated subjects)
Arm/Group | Aripiprazole
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (10.89)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 22
Region of Enrollment [Number; unit: participants]
  Japan | 40

OUTCOME MEASURES:

1. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: Mean change from baseline (Day 1) to endpoint in the YMRS total score
  YMRS is composed of 11 evaluation items with 5 rating levels each. Items rated on a scale of 0 to 4 (comprising 5 rating levels of one point each) are 1) elevated mood, 2) increased motor activity/energy, 3) sexual interest, 4) sleep, 7) language-thought disorder, 10) appearance, and 11) insight. Items rated on a scale of 0 to 8 (comprising 5 rating levels of two points each) are 5) irritability, 6) speech (rate and amount), 8) content, and 9) disruptive-aggressive behavior.
  Total score range is 0 to 60, and the higher value represents worsen.
Time Frame: Day 1 and Day 168 or time of discontinuation
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 40
scores on a scale | -18.8 (9.86)

2. Secondary Outcome: Clinical Global Impression - Bipolar Version (CGI-BP) Sevirity of Illness Score (Mania)
Description: Mean change from baseline (Day 1) to endpoint in Clinical Global Impression -Bipolar Version (CGI-BP) severity of illness score (mania)
  The severity of manic symptoms on a scale of 1 (normal, not ill) to 7 (very severely ill)
Time Frame: Day 1 and Daty 168 or time of discontinuation
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 40
scores on a scale | -2.6 (1.50)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 4/41
Other Adverse Events (participants affected / at risk) | 35/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=41)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1)
Bipolar I Disorder (Psychiatric disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=41)
Nausea (Gastrointestinal disorders) | 9 (9)
Salivary Hypersecretion (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 5 (10)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (8)
Blood Creatine Phosphokinase Increased (Investigations) | 7 (9)
Weight Increased (Investigations) | 7 (7)
Blood Prolactin Decreased (Investigations) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Akathisia (Nervous system disorders) | 18 (20)
Somnolence (Nervous system disorders) | 14 (16)
Tremor (Nervous system disorders) | 9 (10)
Bradykinesia (Nervous system disorders) | 6 (7)
Headache (Nervous system disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 6 (6)
Blister (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No